CLINICAL TRIAL: NCT05403645
Title: Comparison of Exercise Therapy Vs Mobilization With Movement Among Patients With Knee Osteoarthritis in Household Females
Brief Title: Comparison of Exercise Therapy Vs Mobilization With Movement Among Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/502
Record Dates: First submitted 2022-05-05; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Movement; Exercise

STUDY DESIGN:
Intervention Model Description: this study will help to Compare the effect of Exercise Therapy and Movement With Mobilization among patients with knee osteoarthritis in household females
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement With Mobilization among patients with knee osteoarthritis in household females (Experimental): using the techniques of Movement With Mobilization among patients with knee osteoarthritis in household females
  Interventions: Diagnostic Test: Movement With Mobilization
- Exercise Therapy among patients with knee osteoarthritis in household females (Experimental): using the techniques of Exercise Therapy among patients with knee osteoarthritis in household females
  Interventions: Diagnostic Test: Exercise Therapy

INTERVENTIONS:
Diagnostic Test: Movement With Mobilization — with the help of Movement With Mobilization technique
  Arms: Movement With Mobilization among patients with knee osteoarthritis in household females
Diagnostic Test: Exercise Therapy — with the help of Exercise Therapy technique
  Arms: Exercise Therapy among patients with knee osteoarthritis in household females

SUMMARY:
Comparison of exercise therapy Vs mobilization with movement among patients with knee osteoarthritis in household females

DETAILED DESCRIPTION:
To determine the effect of exercise therapy and mulligan*s mobilization with movement techniques on pain and difficulty in performing ADLs with knee OA in household females.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age group of 40-60 included in this study.
* History of knee osteoarthritis, with grade I or II.
* No impairment in other body parts.
* Patients already diagnosed with osteoarthritis by orthopedic surgeon.

Exclusion Criteria:

* Patients with communication problems
* Patients with a history of previous stroke or other neurological diseases or disorders.
* Patients with inflammation.
* Patients who had undergone any surgery.
* Infection or dermatological conditions.
* cardiovascular problems (unstable angina, recent myocardial infarction within the last three months, congestive heart failure, significant heart valve dysfunction etc).

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Exercise Therapy | 6 Months
  intervention in 28 participants which Includeds 3 stretching exercises and 3 strengthening exercises for muscles of knee. Perform each exercise daily for a minimum of 15 seconds for 4 times. The strengthening exercises were also performs daily and each exercise was repeated for 10 times in 3 sets. Pain Visual Analogue Scale(0 for no pain, 10 for maximum pain) & Numerical Pain Rating Scale. used to messure the pain before and after the exercise therapy to acess changes.

SECONDARY OUTCOMES:
Movement With Mobilization | 6 Months
  intervention in 28 participants in which Movement With Mobilization medial glide Movement With Mobilization and medial rotation glide MWM in weight bearing and non-weight positions. MCMASTER OSTEOARTHRITIS INDEX (WOMAC) Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No